CLINICAL TRIAL: NCT03596203
Title: TransCutaneous Magnetic Stimulation (TCMS) for the Treatment of Foot Pain Caused By Diabetic Neuropathy
Brief Title: TCMS for the Treatment of Foot Pain Caused By Diabetic Neuropathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Kashif Munir, Associate Professor, University of Maryland, Baltimore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HP-00081137
Record Dates: First submitted 2018-07-03; First posted 2018-07-23 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Treatment group (Experimental)
  Interventions: Device: TransCutaneous Magnetic Stimulator (TCMS)

INTERVENTIONS:
Device: TransCutaneous Magnetic Stimulator (TCMS) — TCMS coils which are connected to feet and pulse generator. The generator will then be turned on to deliver 50 pulses at a pulse period of 6 seconds and at a pulse intensity of 100% to the bottom of the foot with the TCMS coil.

SUMMARY:
The study will evaluate whether an experimental medical device that emits a series of brief, intense magnetic pulse will relieve foot pain from Diabetic Neuropathy (DN). The United States Food and Drug Administration (FDA) has approved a similar device for treatment of migraine headaches, but this type of device has not been studied for the treatment of DN.

DETAILED DESCRIPTION:
The study will evaluate whether an experimental medical device that emits a series of brief, intense magnetic pulse will relieve foot pain from Diabetic Neuropathy (DN). The United States Food and Drug Administration (FDA) has approved a similar device for treatment of migraine headaches, but this type of device has not been studied for the treatment of DN. No significant adverse reactions or side effects have been reported from the use of magnetic stimulation for the headache treatment. Some patients who have migraine headaches have excellent pain relief with the magnetic treatment even if they did not get pain relief using medications.

The investigators do not know whether this magnetic treatment will relieve the foot pain caused by diabetic neuropathy, so they will test this by applying 50 strong magnet pulses to the painful area of each foot. This procedure will be repeated onto three parts of each foot. First onto the bottom of the foot, then the top of the foot and then the back of the foot including a portion of the ankle. The effect on pain in each foot while walking for about 10 steps will be recorded before the study begins and periodically for 28 days. This testing will provide data as to any improvement in pain relief. If the participants' reported pain is reduced as a result of the magnetic treatment, then the magnetic pulses will have shown that they have reduced the pain. Additional studies will be needed to further investigate this treatment and to determine how to obtain statistically significant data as to whether this therapy reduces the foot pain caused by diabetic neuropathy.

One side effect of this treatment may be some muscular jerking of the foot or the leg during the application of the magnetic pulses. This jerking will last only during the treatment and will not be painful or harmful.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years of age.
2. Prescription pharmacologic treatment is insufficient for treatment of pain.
3. Pain duration of more than one months.
4. Pain occurs daily.
5. Chronic DN associated pain that is located in bilateral feet and is not explained by a central anatomic nerve compression and can clearly be correlated with that patient's history of diabetes.
6. Pain intensity ≥ 5 in each foot at the time of enrollment.

Exclusion Criteria:

1. Life expectancy ≤ 6 months.
2. Oral pain medication doses or active ingredient has changed significantly in the prior 2 weeks.
3. Inability to walk at least 10 steps (with or without a cane) before and after having to sit in a chair.
4. Another pain condition that might confound results (e.g., neuropathy from cancer chemotherapy).
5. Inability to undergo study assessments or complete questionnaires independently.
6. Active psychological co-morbidities (i.e., uncontrolled schizophrenia)
7. Currently using an opioid medication for the treatment of foot pain.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-07-30 (Actual)

PRIMARY OUTCOMES:
Pain level | 1 to 28 days
  Numeric Pain Rating Scale, 0-10 with 0 being no pain, and 10 being worst pain ever experienced

SECONDARY OUTCOMES:
Functional status and Patient satisfaction with treatment | 1 to 28 days
  Descriptive Questionnaire to asses whether participant has improved functional status, such as ability to walk and whether participant is satisfied with treatment
Changes in pain medication | 1 to 28 days
  Assessment of pain medications taken by participant prior to treatment and 28 days after treatment to deteremine if any of pain medications were increased, decreased or eliminated after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Kashif Munir, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Center for Diabetes and Endocrinology, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rao VP, Kim YK, Ghazi A, Park JY, Munir KM. Efficacy of recurrent transcutaneous magnetic stimulation in the treatment of diabetic peripheral neuropathy: Multicenter randomized trial. Pain Pract. 2023 Nov;23(8):914-921. doi: 10.1111/papr.13269. Epub 2023 Jul 3. PMID 37395169
- [Derived] Rao VP, Satyarengga M, Lamos EM, Munir KM. The Use of Transcutaneous Magnetic Stimulation to Treat Painful Diabetic Neuropathy. J Diabetes Sci Technol. 2021 Nov;15(6):1406-1407. doi: 10.1177/19322968211026943. Epub 2021 Jul 3. No abstract available. PMID 34218718